CLINICAL TRIAL: NCT01056575
Title: An Open Label Balanced Study in Healthy Subjects to Evaluate the Potential for Cytochrome P 450 3A4 Induction by Oral OC000459 Using Oral Midazolam as a Probe
Brief Title: Study to Evaluate the Potential for Interaction Between OC000459 and CYP 450 3A4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Dr C Mike Perkins, Oxagen Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OC000459/014/09
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OC000459 (Experimental)
  Interventions: Drug: OC000459

INTERVENTIONS:
Drug: OC000459 — OC000459 100mg tablet, twice daily

SUMMARY:
This will be an open label, sequential study of midazolam (dose 5 mg orally) followed by midazolam (5 mg orally) given after dosing with OC000459 100 mg twice daily for 6.5 days. Twenty subjects will be included to ensure at least 16 subjects with analysable PK data. PK sampling for midazolam and 4-hydroxymidazolam plasma concentrations will continue for up to and including 24 hours after dosing with midazolam on both occasions.

ELIGIBILITY:
Inclusion Criteria:

* Judged to be in good health at screening (blood tests, physical examination, medical history)

Exclusion Criteria:

* Evidence of a clinically significant underlying medical condition that in the opinion of the Investigator would represent a risk to study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Ratio of exposure of midazolam and 4-hydroxymidazolam (without/with exposure to OC000459) as measured by plasma AUC0-t and Cmax for midazolam and its active metabolite 4-hydroxymidazolam. | 6.5 days

SECONDARY OUTCOMES:
Additional PK parameters of midazolam and its active metabolite 4-hydroxymidazolam | 6.5 days
Safety and tolerability of OC000459 | 6.5 days

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, Dr, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom